CLINICAL TRIAL: NCT06962605
Title: Acute Effects of Intermittent vs. Continuous Running Exercise on Physiological and Metabolic Responses
Brief Title: Effects of Intermittent Running on Metabolic Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Normal University (Other)
Responsible Party: Principal Investigator, Yung-Chih Chen, Principal Investigator, National Taiwan Normal University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 202502HM010
Record Dates: First submitted 2025-04-22; First posted 2025-05-08 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Metabolic Regulation; Energy Expenditure
Keywords: Intermittent running; Energy expenditure

STUDY DESIGN:
Intervention Model Description: Participants will be asked to perform 4 trials in a randomized-crossover design (1) moderate-intensity continuous running (MICE: 60% V̇O2max), (2) 5-minute interval running (5MIN; 50% and 70% V̇O2max), (3) 2-minute interval running (2MIN; 50% and 70% V̇O2max).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Moderate-intensity continuous running (MICE: 60% V̇O2max) (Experimental): Exercise
  Interventions: Behavioral: Moderate-intensity continuous running (MICE: 60% V̇O2max)
- 5-minute interval running (5MIN) (Experimental): Exercise
  Interventions: Behavioral: 5-minute interval running (5MIN)
- 2-minute interval running (2MIN) (Experimental): Exercise
  Interventions: Behavioral: 2-minute interval running (2MIN)

INTERVENTIONS:
Behavioral: Moderate-intensity continuous running (MICE: 60% V̇O2max) — Participants run continuously for 40 minutes at moderate intensity (60-65% V̇O2max)
  Arms: Moderate-intensity continuous running (MICE: 60% V̇O2max)
Behavioral: 5-minute interval running (5MIN) — Participants run for 40 minutes at average moderate intensity with 5-minutes slow and fast cycles where speed is increased and decreased by 20%.
  Arms: 5-minute interval running (5MIN)
Behavioral: 2-minute interval running (2MIN) — Participants run for 40 minutes at average moderate intensity with 2-minutes slow and fast cycles where speed is increased and decreased by 20%.
  Arms: 2-minute interval running (2MIN)

SUMMARY:
The purpose of this study is to investigate the suitability of intermittent exercise of long and short intervals at lower intensities than HIIE on energy expenditure during and post-exercise compared to MICE, as well as determine whether similar or greater effects can be achieved for glycemic control in recreationally active adults.

DETAILED DESCRIPTION:
The same procedure will be repeated for all trials: Participants will be asked to perform 3 trials in a randomized-crossover design [moderate-intensity continuous running (MICE: 60% V̇O2max), 5-minute interval running (5MIN; 50% and 70% V̇O2max), 2-minute interval running (2MIN; 50% and 70% V̇O2max)]. All trials will be separated by at least 4 days wash-out and less than 14 days between trials to ensure complete rest.

Sensors for measuring muscle oxygen (10 cm proximal to the mid-patella, and 2 cm lateral) will be placed on the rectus femoris muscle and 15 min resting metabolic rate was measured. After baseline measurements, participants warm-up for 3 minutes with fixed walking intensity (i.e., 5 km/h) followed by 40 minutes running. Immediately after the running, participants return to a seated position for 30 minutes post-exercise measurements (EPOC).

During the EPOC and resting metabolic rate (RMR) measurement participants will sit in a comfortable position and need to limit fidgeting, thus allowed only to watch TV or videos on their phone. Participants will be wheeled to the bathroom if needed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy recreationally active men
* BMI between 18.5-27 kg/m2
* Aged between 20 to 45 years
* Regular exercise (3 times per week and longer than 3 months) with cardio exercise longer than 30 minutes at least once a week
* Weight stable for more than 3 months (no change in weight +/- 3%)
* Non-shift workers and sleep at least 6.5-9 hours for the past 3 months
* Non-smoker

Exclusion Criteria:

* having any cardiovascular, metabolic or pulmonary disease (angina pectoris or uncontrolled arrhythmias)
* suffering from infectious contagious diseases,
* using medications that could affect metabolic responses (including anti-inflammatory medications)
* smoking
* heavy alcohol intake (more than 4 drinks on any day or more than 14 drinks a week).
* undergoing special diets (e.g., intermittent fasting and/or ketogenic diets)

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 16 (Estimated)
Dates: Start 2025-06-21 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Total energy expenditure | 70 minutes
  Changes in total energy expenditure during 40-minutes running and 30 minutes of EPOC
Substrate utilisation | 70 minutes
  Changes in substrate utilisation during 40-minutes running and 30 minutes of EPOC

SECONDARY OUTCOMES:
Muscle oxygen saturation | 70 minutes
  Changes in muscle oxygen during 40 minutes running and 30 minutes EPOC
Subjective appetite sensation | 70 minutes
  Changes in subjective feeling of appetite using 0-100 mm scale (e.g., hunger and satisfaction) during trials

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan Normal University, Taipei, Taiwan